CLINICAL TRIAL: NCT00347542
Title: A Double Blind Randomized Control Trial to Study the Effect of Vitamin D Supplementation on Peripheral Insulin Sensitivity in Centrally Obese Men
Brief Title: A Trial to Study the Effect of Vitamin D Supplementation on Glucose and Insulin Metabolism in Centrally Obese Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sitaram Bhartia Institute of Science and Research (Other)
Responsible Party: Principal Investigator, Dr Jitender Nagpal, Dr Jitender Nagpal, Sitaram Bhartia Institute of Science and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SBISR/2006/03
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2013-06-03 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent; Obesity
Keywords: Vitamin D; Diabetes; Insulin sensitivity; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Insulin Resistance | interventions — Vitamin D

INTERVENTIONS:
Drug: Vitamin D

SUMMARY:
The purpose of the study is to evaluate the change in glucose and insulin metabolism(early markers for development of diabetes) after 6 weeks of weekly Vitamin D supplementation. As vitamin D has been reported to be associated with lipid levels, CRP and blood pressure , we will also be measuring the changes in these variables.

DETAILED DESCRIPTION:
Accumulating evidence suggests that serum Vitamin D levels may be inversely related to the prevalence of diabetes, to the concentration of glucose , insulin resistance and metabolic syndrome.These results have been replicated in patients at risk for diabetes with documentation of impairment in insulin secretion in Vitamin D deficient subjects. Therefore, vitamin D could be implicated in the pathogenesis of type 2 diabetes, by affecting either insulin sensitivity or ß cell function, or both. However, there is paucity of literature on the effect of Vitamin D supplementation on insulin resistance or glucose metabolism. As vitamin D has been reported to be associated with lipid levels, CRP and blood pressure , we will also be measuring the changes in these variables.

ELIGIBILITY:
Inclusion Criteria:

* Male
* ≥35 years of age
* Waist circumference ≥78 cm

Exclusion Criteria:

* Diabetic- Fasting Blood Sugar >126 mg/dl or on anti-diabetic medication
* BP>140/90 or on anti-hypertensive medication
* Receiving Vitamin D or calcium supplementation
* Chronic disease-renal/hepatic/malignancy/gastrointestinal
* On any medication within the last one month which could potentially influence insulin secretion, insulin sensitivity, Vitamin D or Calcium metabolism
* Febrile illness or infective morbidity in the past 10 days
* Past history of nephrolithiasis

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-07; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Insulin Sensitivity (OGIS)

SECONDARY OUTCOMES:
Lipid profile
CRP
ApoA1
ApoB
Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Jitendra N Pande, MD, Principal Investigator — Sitaram Bhartia Institute of Science and Research; Jitender Nagpal, MD, Principal Investigator — Sitaram Bhartia Institute of Science and Research; Anupama Singh, MD, Study Chair — Sitaram Bhartia Institute of Science and Research; Abhishek Bhartia, ME, Study Director — Sitaram Bhartia Institute of Science and Research
Locations (1):
- Sitaram Bhartia Institute of Science and Research, New Delhi, National Capital Territory of Delhi, India